CLINICAL TRIAL: NCT05041127
Title: A Phase II Trial of Cetuximab for Patients With Advanced or Metastatic Chordoma
Brief Title: Cetuximab for the Treatment of Advanced Unresectable or Metastatic Chordoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0217; NCI-2020-14259 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0217 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Chordoma; Metastatic Chordoma; Unresectable Chordoma
MeSH Terms: conditions — Chordoma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cetuximab) (Experimental): Patients receive cetuximab IV over 60-120 minutes QW in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This is a multicenter, single arm, phase 2 study designed to evaluate the efficacy and safety of cetuximab for the treatment of advanced (unresectable)/metastatic, chordoma. The target patient population will be any chordoma patient 18 years of age with locally unresectable disease or metastatic disease.

DETAILED DESCRIPTION:
Primary Objective:

• To evaluate the efficacy of cetuximab in patients with advanced (unresectable) or metastatic, chordoma based on response rate according to RECIST1.1.

Secondary Objectives:

* To evaluate response rate according to Choi criteria
* To evaluate the safety and tolerability of cetuximab for chordoma patients
* To evaluate the progression-free survival (median, at 24 weeks, and 52 weeks) and to determine the overall survival (median).
* To evaluate the ratio of PFS on study compared to PFS from prior treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of chordoma which is advanced (unresectable) and/or metastatic
* ECOG Performance Status of ≤ 2
* At least one site of measurable disease on x-ray/CT/MRI and/or PET/CT scan as defined by RECIST 1.1 criteria. Baseline imaging must be performed within 30 days of Day 1 of study.
* Adequate organ function within 28 days of Day 1 of study defined as:
* The patient has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥ 1000/µL, hemoglobin ≥ 9 g/dL (5.58 mmol/L), and platelets ≥ 100,000/µL
* The patient has adequate hepatic function as defined by a total bilirubin ≤1.5 mg/dL (25.65 μmol/L) (NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper Page 26 limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases).
* The patient has adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed). 3.1.6 Patients may have any prior line of therapy, but there should a washout period of at least 3 weeks from any systemic therapy (small molecule/targeted agents, immunotherapies) and/or radiation therapy.
* Patients should be completely recovered from any reversible toxicities associated with any prior therapies.
* There should be access of archival tumor tissue for central pathology review, or a new tumor related biopsy should be considered within acceptable risk to the patient.
* Patients must have no prior history of use of an EGFR inhibitor for treatment of their chordoma
* Because the teratogenicity of cetuximab is not known, the patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative serum pregnancy test ≤ seven days prior to Day 1 of study.
* Life expectancy of > 3 months

Exclusion Criteria:

* Prior use of an EGFR inhibitor for treatment of their chordoma
* Non-metastatic, resectable disease
* No measurable disease according to RECIST 1.1
* Life expectancy of less than 3 months
* Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured.
* Concomitant participation to another clinical trial with active agent during the study (concomitant non-interventional study will be allowed) Page 27
* Patients who have a history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab, red meat allergy, or tick bite history
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* The patient has clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency.
* The patient has uncontrolled or poorly-controlled hypertension (>180 mmHg systolic or > 130 mmHg diastolic.
* Major surgery within 4 weeks prior to Day 1 of study or who have not recovered adequately from prior surgery
* Patients who have received wide field radiotherapy ≤ 3 weeks or limited field radiation for palliation < 3 weeks prior to Day 1 of study or who have not recovered adequately from side effects of such therapy
* Patients who have received any prior systemic therapy < 3 weeks prior to Day 1 of study or have not recovered adequately from toxicities to the baseline.
* Women who are pregnant or nursing/breastfeeding.
* Inability to comply with protocol required procedures such as Medical, psychiatric, cognitive or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | through study completion, an average of 1 year
  Measured by Response Evaluation Criteria in Solid Tumors 1.1. Will be estimated based on a binomial portion expressed as percentage with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Conley, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT05041127/ICF_000.pdf